CLINICAL TRIAL: NCT01748981
Title: Cardiorespiratory Fitness and Effect of Training After Lung Cancer Surgery. A Randomized Controlled Trial
Brief Title: Fitness, Activity and Lung Cancer Study
Acronym: FALC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian School of Sport Sciences (Other); University Hospital, Akershus (Other); Vestre Viken Hospital Trust (Other)
Responsible Party: Principal Investigator, Elisabeth Edvardsen, Prinsipal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: FALC-2010-OUSNIH
Record Dates: First submitted 2011-08-08; First posted 2012-12-13 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Lung Cancer
Keywords: Pulmonary function; Maximal oxygen uptake; Cardiorespiratory fitness; High-intensity training; Surgery
MeSH Terms: conditions — Lung Neoplasms | interventions — Physical Conditioning, Human

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physical training (Other): Exercise intervention.
  Interventions: Other: Physical training
- As usual (Other): Controls
  Interventions: Other: As usual

INTERVENTIONS:
Other: Physical training — Physical training three times a week for 20 week including endurance and strength training compare to the "as usual" group as controls
  Arms: Physical training
Other: As usual — Controls, not training
  Arms: As usual

SUMMARY:
The purpose of the study is to investigate the change in pulmonary function and exercise capacity in lung cancer patients after pulmonary resection. Furthermore, to study the effect of training on aerobic capacity, muscular strength, morbidity and survival. Physical activity level by accelerometers, body composition by DXA and quality of life will also be reported.

DETAILED DESCRIPTION:
Five year after surgery, all included patients will be reinvited to undergo a fourth health excame to study the long-term effects of exercise training on physical fitness, morbidity and survival.

ELIGIBILITY:
Inclusion Criteria:

* Non smal cell lung cancer
* Patient living in Oslo or Akershus county and accepted for lung cancer surgery at Oslo University hospital and Akershus University hospital
* were able to read and speak Norwegian

Exclusion Criteria:

* Mental incompetence or physical disability that makes it difficult to walk on a treadmill
* Treatment or medical complications affecting ability to participate in an exercise group
* > 79 years

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-06-20 (Actual)

PRIMARY OUTCOMES:
Change in Maximal oxygen uptake (VO2max) from baseline | An expected average of two weeks before surgery (baseline), four to six weeks after surgery, after six months and after 5 years
  Change in VO2max from before to after surgery to measure the effect of surgery, and after six months to measure the effect of high-intensity training intervention, and after five years to study long-term effects

SECONDARY OUTCOMES:
Change in Pulmonary function from baseline | Pulmonary function is measured three times; an expected average of two weeks before surgery, four to six weeks after surgery, after after six months and after five years.
  Change in pulmonary function from before to after surgery and after the intervention

OTHER OUTCOMES:
DXA scan | An expected average of two weeks before surgery, four to six weeks after surgery, after six months and after five years
  Change in body composition from before to after surgery and after the intervention
Quality of life | Measured three times: An expected average of two weeks before surgery, four to six weeks after surgery, after six months and after five years
  Change in quality of life from before to after surgery and after the intervention
Physical activity | Measured three times: six weeks after surgery, after six months and after five years
  Physical activity will be objectively measured by accelerometers for seven consecutive days to determine change in activity level after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Edvardsen, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Edvardsen E, Skjonsberg OH, Holme I, Nordsletten L, Borchsenius F, Anderssen SA. High-intensity training following lung cancer surgery: a randomised controlled trial. Thorax. 2015 Mar;70(3):244-50. doi: 10.1136/thoraxjnl-2014-205944. Epub 2014 Oct 16. PMID 25323620
- [Derived] Edvardsen E, Anderssen SA, Borchsenius F, Skjonsberg OH. Reduction in cardiorespiratory fitness after lung resection is not related to the number of lung segments removed. BMJ Open Sport Exerc Med. 2015 Oct 5;1(1):e000032. doi: 10.1136/bmjsem-2015-000032. eCollection 2015. PMID 27900127